CLINICAL TRIAL: NCT07218900
Title: A Phase II, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Effect of AZD0780 in Combination With Rosuvastatin on Low Density Lipoprotein Cholesterol in Participants With Dyslipidaemia (LAZURE)
Brief Title: A Study to Investigate the Effect of AZD0780 Tablets in Combination With Rosuvastatin Tablets on Low Density Lipoprotein Cholesterol Levels (LDL-C) in Adult Participants With Dyslipidaemia
Acronym: LAZURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ-RU-00013
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Dyslipidaemia
Keywords: AZD0780; Dyslipidaemia; Low-Density Lipoprotein Cholesterol
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Multi-centre, randomised, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD0780 +Rosuvastatin (Experimental): Participants will receive Rosuvastatin for 28 days. Then receive AZD0780 on top of rosuvastatin, administered orally for 12 weeks
  Interventions: Drug: AZD0780; Drug: Rosuvastatin
- Placebo +Rosuvastatin (Placebo Comparator): Participants will receive Rosuvastatin for 28 days. Then receive Placebo on top of rosuvastatin, administered orally for 12 weeks
  Interventions: Drug: Placebo; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Placebo — Administered orally as tablets
  Arms: Placebo +Rosuvastatin
Drug: AZD0780 — Administered orally as tablets
  Arms: AZD0780 +Rosuvastatin
Drug: Rosuvastatin — Administered orally as tablets

SUMMARY:
This is a study to investigate the effect of AZD0780 tablets on low density lipoprotein cholesterol levels (LDL-C) compared with placebo tablets administered in combination with rosuvastatin tablets in adult Russian participants with dyslipidaemia. AZD0780 is a small molecule that reduces the amount of LDL-C in the blood. Placebo will be used for comparison, and neither the participants nor the Investigators will know who is receiving the AZD0780 medication and who is receiving the placebo until the end of study.

The total length of the study for an individual participant will be up to 136 days, including a screening period of up to 14 days, rosuvastatin run-in period of 28 days, treatment with AZD0780 or placebo for 84 days, and a safety follow-up period of 10 days.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group Phase II study to evaluate the effect of AZD0780 on the reduction of LDL-C, as well as its safety and tolerability, compared to placebo. The study drug will be administered orally once daily in addition to rosuvastatin for up to 12 weeks in participants receiving moderate-intensity statin therapy or not receiving any statin therapy. The target population is adults ≥ 18 years of age with LDL-C ≥ 55 mg/dL and history of clinical Atherosclerotic cardiovascular disease (ASCVD) or ≥ 70 mg/dL and at risk for a first ASCVD event.

The study will be conducted at approximately 11 centres in Russia.

The screening period is up to 14 days, starts at the date of signed informed consent, and ends on the day before the randomisation visit. Participants who meet all screening inclusion criteria and do not meet any exclusion criterion will enter a run-in period with rosuvastatin for 28 days before randomisation. Participants will be randomised in a 1:1 ratio to either AZD0780 or placebo for a treatment period of 12 weeks and a 10-day safety follow-up. Those randomised to the AZD0780 group will receive AZD0780 orally once daily in addition to rosuvastatin during the treatment period, while those in the placebo group will receive matching placebo in addition to rosuvastatin. The study will include approximately 76 randomised participants.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of signing the ICF
* History of clinical Atherosclerotic cardiovascular disease (ASCVD) or at risk for a first ASCVD event:

  1. Clinical ASCVD is defined as MI, stable or unstable angina, coronary or other arterial revascularisation, ischaemic stroke, or peripheral artery disease.
  2. A participant is considered at risk for a first ASCVD event if the participant has one or more of the following conditions: atherosclerotic vascular disease (≥ 50% stenosis in ≥ 2 coronary artery territories or in ≥ 2 vascular beds [coronary, carotid, lower extremity], diagnosed by any imaging modality), diabetes mellitus, hypertension, cigarette smoking, chronic kidney disease (moderate to severe stage), or obesity. Investigators can also use the ACC/AHA or ESC or national clinical guidelines for risk assessment to identify participants with at least moderate risk for ASCVD.
* Fasting serum LDL-C by central laboratory at screening as follows: LDL-C ≥ 55 mg/dL (≥ 1.4 mmol/L) in participants with clinical ASCVD or ≥ 70 mg/dL (≥ 1.8 mmol/L) in participants without clinical ASCVD but at risk for a first ASCVD event
* Participants should meet 1 of the following before screening:

  1. On a stable dose of Lipid-lowering therapy (LLTs) including moderate statins.
  2. On a stable dose of LLTs without any statins (either have been previously treated or be statins treatment naïve).
  3. Not received treatment with any LLTs (either have been previously treated or be LLTs treatment naïve).

Exclusion Criteria:

* Homozygous familial hypercholesterolaemia, known diagnosis of heterozygous familial hypercholesterolaemia (HeFH), LDL apheresis or plasma apheresis within 12 months prior to screening, or any other underlying known disease or condition that may interfere with interpretation of the clinical study results as judged by the Investigator.
* Any of the following laboratory values at screening:

  1. Calculated eGFR < 15 mL/min/1.73 m2
  2. AST or ALT > 3 × ULN
  3. TBL > 2 × ULN (except for patients with Gilberts syndrome, where TBL 3 × ULN is acceptable provided direct bilirubin < 1.5 × ULN)
  4. Fasting triglycerides ≥ 400 mg/dL (≥ 4.52 mmol/L)
  5. Creatine kinase > 5 × ULN
  6. Urine albumin-to-creatinine ratio ≥ 500 mg/g
* Uncontrolled type 2 diabetes mellitus defined as HbA1C ≥ 9.5% at screening
* Inadequately treated hypothyroidism defined as TSH > 1.5 ULN at screening or participants whose thyroid replacement therapy was initiated or modified within the last 3 months prior to screening
* Use of mipomersen or lomitapide (cholesterol-lowering medications) within 12 months prior to screening or planned use during the study.
* Use of gemfibrozil within 1 week prior to screening or planned use during the study.
* Use of PCSK-9 inhibitors: evolocumab/alirocumab within 12 weeks of the screening visit or planned use during the study or inclisiran within 18 months of the screening visit or planned use during the study. Any other approved PCSK-9 inhibitor use within 5 half-lives prior to the screening visit or planned use during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Relative change in Low-density lipoprotein cholesterol (LDL-C) from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on LDL-C at 12 weeks

SECONDARY OUTCOMES:
Indicator for LDL-C < 70 mg/dL (< 1.8 mmol/L) at 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on the probability of LDL-C < 70 mg/dL at 12 weeks in patients with baseline LDL-C ≥ 70 mg/dL
Indicator for LDL-C < 55 mg/dL (< 1.4 mmol/L) at 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on the probability of LDL-C < 55 mg/dL at 12 weeks
Relative change in Apolipoprotein (Apo) B from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on Apo B at 12 weeks
Relative change in non-high-density lipoprotein cholesterol (non-HDL-C) from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on non-HDL-C at 12 weeks
Relative change in total cholesterol from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on total cholesterol at 12 weeks
Relative change in lipoprotein(a) (Lp[a]) from baseline to 12 weeks | Baseline - 12 weeks
  To compare the effect of treatment with AZD0780 versus placebo on Lp[a] at 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Research Site, Aramil
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at : https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home